CLINICAL TRIAL: NCT03559764
Title: Clinical Study on the Safety and Efficacy of Anti-BCMA CAR T Cells With Relapsed and Refractory Multiple Myeloma
Brief Title: Study of BCMA CAR-T in Multiple Myeloma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allife Medical Science and Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCMA CAR T-HNRM-01
Record Dates: First submitted 2018-05-08; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Relapsed and Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-BCMA CAR T cells (Experimental): Total dose of 0.5-6 millions /kg cells will be administered at day -2, day -1 and day 0 by split dose (30%, 30% and 40% respectively).
  Interventions: Biological: Anti-BCMA CAR T cells

INTERVENTIONS:
Biological: Anti-BCMA CAR T cells — Transparent colorless or slightly yellow liquid

SUMMARY:
This is a single centre、single arm、open-label，to investigate the safety and efficacy of anti-BCMA CAR T cells in patients with Relapsed and Refractory multiple myeloma.

DETAILED DESCRIPTION:
Multiple myeloma（MM） is one of the most common malignant diseases in the blood system.There is still no cure for the disease which only control the development of the disease in various ways.CAR - T cells was taken in the form of genetic modification, and specific identified target antigen monoclonal antibody of single variable region (scFv) expression in T cell surface, and coupled with the activation of intracellular proliferation signal domain. The study will follow a 3 + 3 design of dose-escalating cohorts. After a patient enrolls,leukapheresis will be performed to obtain peripheral blood mononuclear cells which will be sent to a manufacturing site to produce anti- BCMA CAR T cells. The cells will then be returned to the investigational site and, after a standard chemotherapy based conditioning regimen, will be administered to the patient. Treated patients will undergo serial measurements of safety, tolerability and response.

In order to lay a foundation for the application of relapsed/refractory multiple myeloma patients with CAR-T therapy，objects are refractory/ relapsed patients with multiple myeloma,and plans to into the group of the number of cases in 20 cases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 70 years old (including 18 and 70 years old)
2. BCMA antigen diagnosed by pathology and histological examination was positive
3. ECOG ≤2，and the excepted survival ≥ 3 months
4. Patients with BCMA+ myeloma who received ≥ 1 line of chemoradiotherapy or tumor relapsed
5. The main organs function is good; （1） liver function: ALT/AST<3 times normal value upper limit (ULN) and total bilirubin <34.2 (mol/L); （2） renal function: creatinine <220 mu /L,GFR > 30mL/min; （3） lung function: blood oxygen saturation is greater than 95%; （4） cardiac function: left ventricular ejection fraction (LVEF) is greater than 50%;
6. Platelets > 40 billion/L;
7. Patients without any anti-cancer treatment such as chemotherapy，radiotherapy, immunotherapy（ immunosuppressive drugs ）within 2-4 weeks before, and the treatment-related toxicity reaction ≤1 level prior to enrollment（except low toxicity lose hair for example）
8. Venous channel is unobstructed, which can meet the needs of intravenous drip;
9. Voluntary informed consent is given, agree to follow the trial treatment and visit plan.

Exclusion Criteria:

1. Patients with allergy to large molecules such as antibodies or cytokines;
2. More than 5mg of hormones (except patients with inhaled hormone) were used within 2 to 4 weeks prior enrollment;
3. Patients with severe autoimmune diseases or immunodeficiency diseases;
4. Patients treated with other immune cellular products (DC, CIK, T, NK, and CART products with CD19 or other targets);
5. Patients with uncontrollable infectious disease in the first 4 weeks of treatment;
6. Active hepatitis B DNA > 1000copy/mL/ , hepatitis C positive, (HCV positive resistance, HCV RNA positive);
7. Patients participated in other clinical trials within 6 weeks prior enrollment;
8. Patients with mental illness;
9. Patients with drug abuse/addiction and medical, psychological or social conditions may interfere with the study or evaluate the results of the study;
10. Patients have alcohol dependence;
11. Pregnant or lactating women; Men or women who have a pregnancy plan within a year; The patients cannot guarantee effective contraceptive measures during the trial period;
12. Patients had other conditions that were not appropriate for the group determined by the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
The safety of CAR T is evaluated to determine if CRS occurred | Day 3-Year 2 after injection
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment